CLINICAL TRIAL: NCT04501497
Title: Prospective Multicenter Observational Study of Atezolizumab Combination Therapy in Patients With Unresectable, Advanced and Recurrent Non-small Cell Lung Cancer or Extensive Disease Small Cell Lung Cancer
Brief Title: Prospective Multicenter Observational Study of Atezolizumab Combination Therapy in Lung Cancer (J-TAIL-2)
Status: Completed | Type: Observational
Sponsor: Chugai Pharmaceutical (Industry)
Collaborators: Japan Lung Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: J-TAIL-2
Record Dates: First submitted 2020-08-02; First posted 2020-08-06 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer; Extensive Disease Small Cell Lung Cancer
Keywords: Atezolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSCLC cohort (N=800): Patients with locally advanced or metastatic non-small cell lung cancer who are planning to provide Atezolizumab combination thearapy as the most ppropriate medical care
- ED-SCLC cohort (N=400): Patients with extensive disease small cell lung cancer who are planning to provide Atezolizumab combination thearapy as the most ppropriate medical care

SUMMARY:
This is a multi-center observational study of atezolizumab combination therapy in patients with unresectable, advanced and recurrent non-small cell lung cancer(NSCLC) or extensive disease small cell lung cancer(ED-SCLC). 800 patients in NSCLC cohort and 400 patients in ED-SCLC cohort will be enrolled in this trial to assess the efficacy and safety of this combination.

DETAILED DESCRIPTION:
Primary endpoint: 12 months OS, Secondary endpoints: Overall Survival(OS), 6 months survival rate(6mo OS), 12 months survival rate(12mo OS), Progression-Free Survival(PFS), Time to treatment failure (TTF), Objective Response Rate(ORR), Disease Control Rate(DCR), Duration of Response(DOR) ,Safety and Comprehensive geriatric assessment(G8)

ELIGIBILITY:
Inclusion Criteria:

< non-small cell lung cancer cohort>

1. Patients 20 years of age or older at the time of signed consent.
2. Patients with unresectable, advanced and recurrent non-small cell lung cancer.
3. Patients who are scheduled to start atezolizumab combination therapy in clinical practice, based on the atezolizumab package insert and the Optimal Use Promotion Guideline.
4. Patients who signed informed consent form before enrolling the study. The consent from a legally acceptable representative is required for the patients with uncertain capacity of judgments.

<extensive disease small cell lung cancer cohort>

1. Patients 20 years of age or older at the time of signed consent.
2. Patients with extensive disease small cell lung cancer.
3. Patients who are scheduled to start atezolizumab combination therapy in clinical practice, based on the atezolizumab package insert and the Optimal Use Promotion Guideline.
4. Patients who signed informed consent form before enrolling the study. The consent from a legally acceptable representative is required for the patients with uncertain capacity of judgments.

Exclusion Criteria:

< non-small cell lung cancer cohort> (1) Patients who are unsuitable for enrolment into the study by the investigator's judgment.

<extensive disease small cell lung cancer cohort>

(1) Patients who are unsuitable for enrolment into the study by the investigator's judgment.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are planning to provide Atezolizumab combination therapy as the most appropriate medical care for patients and who meet the Eligibility criteria at registration.
Sampling Method: Non-Probability Sample
Enrollment: 1221 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
12 months survival rate | Baseline up to 12 Months
  Percentage of participants alive 12 months after initiation of treatment

SECONDARY OUTCOMES:
Overall Survival | Up to death (up to 3 years)
  OS was defined as the time from the first day of study treatment to death due to any cause
6 moths survival rate | Up to 6 months
  Percentage of participants alive 6 months after initiation of treatment
18 moths survival rate | Up to 18 months
  Percentage of participants alive 18 months after initiation of treatment
Progression-Free Survival(PFS) | Up to disease progression or death whichever occurs first (up to 3 years)
  PFS based on disease status as evaluated by the investigator in accordance with Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (v1.1)
Time to treatment failure (TTF) | Up to 3 years
  TTF was defined as the time from the first day of study treatment to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death
Post-treatment transfer rate | Up to post-treatment is started (up to 3 years)
  Rate of patients who received drug therapy for primary disease after study treatment
Objective Response Rate(ORR) | Up to disease progression or death whichever occurs first (up to 3 years)
  Percentage of participants with objective response as assessed by the investigator according to RECIST v1.1
Duration of Response(DOR) | From date of first objective response up to disease progression or death whichever occurs first (up to 3 years)
  Duration of Response as Assessed by the Investigator According to RECIST v1.1
Disease Control Rate(DCR) | Up to 3 years
  Percentage of patients with controled disease as Assessed by the investigator according to RECIST v1.1
Percentage of Participants with adverse events(Adverse Reactions) | Up to 3 years
  The incidence of worst-grade adverse events on study as graded by NCI-CTCAE v5.0
Comprehensive geriatric assessment (G8) | At baseline
  The G-8 screening tool was developed to identify elderly cancer patients who would benefit from comprehensive geriatric assessment

CONTACTS AND LOCATIONS:
Overall Officials: Akihiko GENMA, Principal Investigator — Nippon Medical School Hospital
Locations (148):
- Japan (148):
  - Akashi Medical Center, Akashi
  - Hyogo Cancer Center, Akashi
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki
  - Asahikawa Medical University Hospital, Asahikawa
  - National Hospital Organization Asahikawa Medical Center, Asahikawa
  - Juntendo University Hospital, Bunkyō City
  - Nippon Medical School Hospital, Bunkyō City
  - Tokyo Medical And Dental University, Medical Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - National Cancer Center Hospital, Chūōku
  - Fujisawa City Hospital, Fujisawa
  - Fukui Prefectural Hospital, Fukui
  - Fukuoka University Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Gifu Prefectural General Medical Center, Gifu
  - National Hospital Organization Okinawa National Hospital, Ginowan
  - Hamamatsu University Hospital, Hamamatsu
  - National Hospital Organization Himeji Medical Center, Himeji
  - Kansai Medical University Hospital, Hirakata
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Aso Iizuka Hospital, Iizuka
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai
  - Japanese Red Cross Ise Hospital, Ise
  - Tokai University Hospital, Isehara
  - Teikyo University Hospital, Itabashi-Ku
  - Itami City Hospital, Itami
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni
  - Shimane University Hospital, Izumo
  - Juntendo University Shizuoka Hospital, Izunokuni
  - Kagawa University Hospital, Kagawa
  - Kagoshima University Hospital, Kagoshima
  - Kameda Medical Center, Kamogawa
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - Kanazawa University Hospital, Kanazawa
  - Ibaraki Prefectural Central Hospital, Kasama
  - Kasukabe Medical Center, Kasukabe
  - Kishiwada City Hospital, Kishiwada
  - Hospital of the University of Occupational and Envioronmental Health, Kitakyushu
  - Japan Community Health care Organization Kyushu Hospital, Kitakyushu
  - Kitakyushu Municipal Medical Center, Kitakyushu
  - Japan Anti-Tuberculosis Association Fukujuji Hospital, Kiyose
  - National Hospital Organization Tokyo National Hospital, Kiyose
  - Kobe City Medical Center General Hospital, Kobe
  - Kobe Minimally Invasive Cancer Center, Kobe
  - Kobe University Hospital, Kobe
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Kōtoku
  - Kurashiki Central Hospital, Kurashiki
  - National Hospital Organization Kure Medical Center and Chugoku Cancer, Kure
  - Kurume University Hospital, Kurume
  - Kyoto City Hospital, Kyoto
  - Kyoto University Hospital, Kyoto
  - Kyoto-Katsura Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Matsusaka Municipal Hospital, Matsusaka
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - National Hospital Organization Tokyo Medical Center, Meguro-Ku
  - The Jikei University Hospital, Minatoku
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki
  - Nagahama City Hospital, Nagahama
  - Aichi Medical University Hospital, Nagakute
  - Nagasaki University Hospital, Nagasaki
  - Aichi Cancer Center, Nagoya
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Nagoya Ekisaikai Hospital, Nagoya
  - Nagoya University Hospital, Nagoya
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Miyagi Cancer Center, Natori
  - Niigata Cancer Center Hospital, Niigata
  - Niigata University Medical and Dental Hospital, Niigata
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Obihiro Kosei Hospital, Obihiro
  - Japanese Red Cross Okayama Hospital, Okayama
  - Kawasaki Medical School General Medical Center, Okayama
  - Okayama Rosai Hospital, Okayama
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Oita Prefectural Hospital, Ōita
  - Kindai University Hospital, Ōsaka-sayama
  - Osaki Citizen Hospital, Ōsaki
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Shiga University of Medical Science Hospital, Ōtsu
  - Saga University Hospital, Saga
  - Kitasato University Hospital, Sagamihara
  - Jichi Medical University Saitama Medical Center, Saitama
  - Saitama medical university International medical Center, Saitama
  - Saitama Prefectural Cancer Center, Saitama
  - Saitama Red Cross Hospital, Saitama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai
  - Hokkaido University Hospital, Sapporo
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - Sapporo Medical University Hospital, Sapporo
  - Teine Keijinkai Hospital, Sapporo
  - Sendai Kousei Hospital, Sendai
  - Tohoku Medical And Pharmaceutical University Hospital, Sendai
  - Tohoku University Hospital, Sendai
  - Japanese Red Cross Medical Center, Shibuya-Ku
  - Jichi Medical University Hospital, Shimotsuke
  - Showa University Hospital, Shinagawa-Ku
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku
  - Keio University Hospital, Shinjuku-Ku
  - Tokyo Medical University Hospital, Shinjuku-Ku
  - Iwate Medical University Hospital, Shiwa-gun
  - Shizuoka Cancer Center, Shizuoka
  - Shizuoka General Hospital, Shizuoka
  - Osaka University Hospital, Suita
  - Saiseikai Suita Hospital, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - JA Toyama Kouseiren Takaoka Hospital, Takaoka
  - Takarazuka City Hospital, Takarazuka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Tenri Hospital, Tenri
  - Dokkyo Medical University Hospital, Tochigi
  - Tokushima Prefectural Central Hospital, Tokushima
  - Tokushima University Hospital, Tokushima
  - Toyama Prefectural Central Hospital, Toyama
  - Fujita Health University Hospital, Toyoake
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka
  - TOYOTA Memorial Hospital, Toyota
  - Ehime University Hospital, Tōon
  - Tsukuba Medical Center Hospital, Tsukuba
  - University of Tsukuba Hospital, Tsukuba
  - National Hospital Organization Yamaguchi-Ube Medical Center, Ube
  - Juntendo University Urayasu Hospital, Urayasu
  - Japanese Red Cross Wakayama Medical Center, Wakayama
  - Wakayama Medical University Hospital, Wakayama
  - Kanagawa Cancer Center, Yokohama
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Yokohama City University Hospital, Yokohama
  - Yokohama Municipal Citizen's Hospital, Yokohama
  - Yokosuka Kyosai Hospital, Yokosuka
  - Tottori University Hospital, Yonago
  - Oita University Hospital, Yufu

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the end of the study